CLINICAL TRIAL: NCT06005519
Title: The Short and Long-term Effects of Low AGE Diet on Individuals With and Without Type 2 Diabetes
Brief Title: The Short and Long-term Effects of Low Advanced Glycation End Product* Diet
Acronym: AGE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University Pendik Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Buğu Usanma Koban, Asst Prof, Marmara University Pendik Training and Research Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 480
Record Dates: First submitted 2023-08-14; First posted 2023-08-22 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: Diabetes Type 2
Keywords: Advanced glycation end products; diabetes; nutrition; diet
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Type 2 diabetes (Other)
  Interventions: Other: low AGE diet education
- healthy participants (Other)
  Interventions: Other: low AGE diet education

INTERVENTIONS:
Other: low AGE diet education — Participants were divided into ten-person groups. Each group was individually invited for a face-to-face meeting where they were provided with a 50-minute low-AGE diet education prepared in accordance with the recommendations of the American Diabetes Association and the Turkish Society of Endocrinology and Metabolism. During the first 20 minutes of the education, a PowerPoint presentation highlighted the importance of choosing plant-based, low-AGE foods and emphasized cooking methods such as boiling, steaming, and preparing meals with added liquids. Participants were advised against frying, roasting, and grilling. Additionally, information was provided on marinade techniques and the use of spices or ingredients such as lemon or vinegar to lower pH in meals. Following the education, participants were given a dietary diary to record their food intake and were asked to self-assess their diet adherence on a scale of 1 to 10 on a weekly basis.

SUMMARY:
The aim of this study was to examine the hypothesis that a diet low in advanced glycation end products (AGE) would provide short and long term improvement in metabolic and inflammatory parameters and serum AGE, Srage, carboxymethyllysine (CML) and methylglyoxal (MG) values in individuals with type 2 diabetes. Specifically, in order to observe the effect of AGE content on the results, diabetic patients who are followed up and who know the principles of low glycaemic index and glycaemic load nutrition suitable for diabetic patients, who do not have additional diseases and who do not smoke were selected.

In recent years, it has been determined that AGE accumulation in the tissue has an effect on the pathophysiology of many diseases such as Alzheimer's disease as well as chronic complications of diabetes. However, the contribution of dietary AGE intake to this pool is controversial. There are studies with conflicting results in the literature on whether a low AGE diet is effective on metabolic and biochemical well-being. In addition, studies investigating the effects of reducing AGE content in the diet of people with no chronic disease are limited.

In this study, the metabolic results of dietary modification in the short term of 2 weeks and in the long term of 3 months are determined. In addition, the results are analysed separately in type 2 diabetic and non-diabetic groups. Thus, the data showing the short and long term metabolic effects of dietary AGE levels for diabetic and non-diabetic patients will contribute to the literature.

DETAILED DESCRIPTION:
The study included 30 volunteers with type 2 diabetes and 30 healthy participants. During the initial interviews, participants were provided with training on low AGE (advanced glycation end-products) dietary principles. In the same session, measurements were taken and recorded for height, body weight, blood pressure, waist and hip circumference, and body fat percentage. Fasting blood glucose, HbA1c, c-peptide, C reactive protein (CRP), insulin, blood lipid levels, 1-5 anhydroglucitol (1-5 AG), AGE, Soluble AGE Receptor (sRAGE) , methylglyoxal (MG) and carboxymethyllysine (CML) levels were measured through blood samples.

Participants were asked to maintain a dietary journal and were followed up through weekly online or face-to-face meetings. They were called in for a follow-up examination 2 weeks and 3 months after the initial interview. Anthropometric measurements and blood tests were repeated.

After the completion of a 3-month follow-up for all participants, measurements from both the short and long term resulting from the low AGE diet were analyzed by comparing them to the initial measurements, both for participants with and without diabetes.

ELIGIBILITY:
Inclusion Criteria:

* To have the competence to adhere to dietary recommendations

Exclusion Criteria:

* Being <18 years old or >65 years old
* Having a history of serious cardiovascular diseases (atrial fibrillation, stroke, ischemic heart disease, peripheral vascular disease, heart failure)
* Having chronic obstructive pulmonary disease
* Smoking
* Having kidney or liver failure
* Having a chronic gastrointestinal disease associated with malabsorption or chronic pancreatitis
* Having a history of rheumatological disease
* Having a history of severe acute illness, malignancy, or alcohol abuse in the last 1 month
* Receiving immunosuppressive treatment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2021-08-30 (Actual)

PRIMARY OUTCOMES:
Change in serum AGE levels in short time period | 14 days
  After a 2-week low AGE diet, a change in serum AGE levels in the diabetic and nondiabetic groups
Change in serum AGE levels in long time period | 90 days
  After a 3 months low AGE diet, a change in serum AGE levels in the diabetic and nondiabetic groups
change in body weight in short time period | 14 days
  After a 2-week low AGE diet,change in body weight (kg) in diabetic and nondiabetic groups
Change in body weight in long time period | 90 days
  After a 3-months low AGE diet, change in body weight (kg) in diabetic and nondiabetic groups
change in body mass index in short time period | 14 days
  After a 2-week low AGE diet,change in body mass index in diabetic and nondiabetic groups
change in body mass index in long time period | 90 days
  After a 3-months low AGE diet, change in body mass index in diabetic and nondiabetic groups
change in waist circumference in short time period | 14 days
  After a 2-week low AGE diet, change in waist circumference (cm) in diabetic and nondiabetic groups
change in waist circumference in long time period | 90 days
  After a 3-months low AGE diet, change in waist circumference (cm) in diabetic and nondiabetic groups
change in hip circumference in short time period | 14 days
  After a 2-week low AGE diet, change in hip circumference (cm) in diabetic and nondiabetic groups
change in hip circumference in long time period | 90 days
  After a 3-months low AGE diet, change in hip circumference (cm) in diabetic and nondiabetic groups
change in body fat percentage in short time period | 14 days
  After a 2-week low AGE diet,change in body fat percentage (%) in diabetic and nondiabetic groups
change in body fat percentage in long time period | 90 days
  After a 3-months low AGE diet,change in body fat percentage (%) in diabetic and nondiabetic groups

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University Istanbul Medical Faculty, Istanbul, Fatih, Turkey (Türkiye)